CLINICAL TRIAL: NCT06821438
Title: PREOPERATIVE TRANSVAGINAL ULTRASOUND VERSUS MAGNETIC RESONANCE IMAGING IN DIAGNOSIS OF LAPAROSCOPICALLY MANAGED PATIENTS WITH DEEP INFILTRATING ENDOMETRIOSIS
Brief Title: TVUS vs MRI Efficacy in Diagnosis of Laparoscopically Managed Patients With DIE
Status: Not yet recruiting | Type: Observational
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Tamer Hosny, Principal investigator Dr Tamer Ahmed Hosny, Alexandria University
Other Study IDs: US vs MRI in DIE
Record Dates: First submitted 2025-01-05; First posted 2025-02-12 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Endometriosis
MeSH Terms: conditions — Endometriosis | interventions — Laparoscopy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Laparoscopy — Endoscopy

SUMMARY:
The purpose of the study is to compare the reliability and accuracy of systematic ultrasonographic scanning using International Deep Endometriosis Analysis group approach versus magnetic resonance imaging (MRI) assessment in diagnosis of patients with deep infiltrative endometriosis in comparison with the intraoperative findings to confirm the accuracy.

DETAILED DESCRIPTION:
Endometriosis is the existence of endometrial glands outside the uterus. About 10%- 12% of women who are menstruating have this benign gynecologic disease with peak age between 25 years and 35 years. However asymptomatic women can develop endometriosis lesions, and half of those suffering from infertility are found to have them. Endometriosis currently poses a significant problem because of its complexity, the range of clinical presentations it might take, and the still unknown physio-pathobiological genesis. There are three types of endometriosis; Deep Infiltrating Endometriosis, ovarian endometrioma, and superficial peritoneal endometriosis.

Deep infiltrating endometriosis is defined as the ectopic growth of endometrial glands and stroma extending more than 5 mm beneath the peritoneal surface. This type needs special and more vigorous management than the other types. It accounts for 15-30% of all the diagnosed endometriosis cases.

Ovarian endometrioma which is defined as "Endometrium-like tissue in the form of ovarian cysts "chocolate cysts". it is found in 2-10% of women in reproductive age and half of women receiving infertility treatment.

Superficial peritoneal endometriosis which is defined as "Endometrium- like tissue lesions involving the peritoneal surface. The lesions can have different appearances and color e.g. clear, black, etc.". It represent 15-50% of diagnosed cases.

This illness can cause crippling pain, infertility, and problems with bowel, sexual, and urine functions. These symptoms can have a major negative impact on a woman's quality of life during her reproductive years.

Because Deep Infiltrating Endometriosis tends to profoundly infiltrate pelvic systems, including several organs, ligaments, blood arteries, and nerves, it might mimic malignant processes despite being benign. Extensive and intricate dissection inside deep pelvic regions is necessary for the complicated excision of Deep Infiltrating Endometriosis in its aggressive form.

Noninvasive imaging modalities such as magnetic resonance imaging and transvaginal sonography are currently available for the diagnosis of Deep Infiltrating Endometriosis.

Regardless of its location, it is crucial to remember that there is significant variation in the stated sensitivity and specificity of transvaginal ultrasound for Deep Infiltrating Endometriosis detection.

The diagnosis of pelvic endometriosis is more accurate when an expert operator does an ultrasonography according to International Deep Endometriosis Analysis approach in addition to a pelvic examination and history.

When a woman has endometriosis, an ultrasound examination is performed to map the location of the disease, determine its severity, and attempt to explain the underlying symptoms before pursuing medication or surgery.

However, discrepancies in examination techniques, ultrasound equipment quality, and operator experience may account for discrepancies in the reported accuracy of the ultrasound diagnosis of Deep Infiltrating Endometriosis across different investigations.

MRI has a great degree of objectivity and the ability to capture pictures in various orientations over a wide field of view. The fusion of many Magnetic Resonance sequences can provide extensive information regarding the sites and histological aspects of endometriosis because of its superior contrast resolution.

The diagnosis is usually made through surgical visualization, ideally laparoscopy, although the recent guidelines from ESHRE suggest that actual imaging modalities for some types of endometriosis could be sufficient in the diagnosis process.

At present, there is no curative treatment for endometriosis, and clinical management of symptoms such as pain occurs through medical and/or surgical treatments .

Medical treatment follows the basic principle of suppression of menstrual cycles, resulting in the reduction in inflammation and blocking the effect of estrogens [Falcone 2018]. Unfortunately, current medical therapies could alleviate symptoms, but they are far from curative treatments and can often lead to side effects that compromise patient compliance.

Surgical treatment aims to remove bulky endometriotic lesions or, in more complex cases, complete excision of the pelvic organs. Neither the medical management nor the surgery turns out to give relief in the long term or is universally acceptable for the patients.

Laparoscopic observation and biopsy are very important in the diagnosis of Deep Infiltrating Endometriosis where the specimens biopsied are sent for histopathological examination for diagnosis of the nature of the lesions and their exact origin.

ELIGIBILITY:
Inclusion Criteria:

* Known patient with Deep Infiltrating Endometriosis affecting ovaries (endometriomas), rectosigmoid , bladder or any type of endometriosis who suffers from chronic pelvic pain, dysmenorrhea, dyspareunia, dyschasia, dysuria or infertility.

Exclusion Criteria:

* Postmenopausal status.
* Women with malignancy or adnexal lesions other than suspected endometrioma.
* Those who were pregnant.
* History of any metallic implants or prosthesis preventing MRI. 5. Virgin cases (No Transvaginal Ultrasound).

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients with Deep Infiltrating Endometriosis affecting ovaries (endometriomas), rectosigmoid , bladder or any type of endometriosis who suffers from chronic pelvic pain, dysmenorrhea, dyspareunia, dyschasia, dysuria or infertility. All cases included were subjected to the following: History taking, analysis of complaint, physical examination , transvaginal sonography, MRI and laparoscopy. These are done after informed written consents.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-02 (Estimated); Primary Completion 2025-04 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
TRANSVAGINAL ULTRASOUND VERSUS MAGNETIC RESONANCE IMAGING IN DIAGNOSIS OF LAPAROSCOPICALLY MANAGED PATIENTS WITH DEEP INFILTRATING ENDOMETRIOSIS | Baseline
  The purpose of the study is to compare the reliability and accuracy of systematic ultrasonographic scanning using International Deep Endometriosis Analysis group approach versus magnetic resonance imaging (MRI) assessment in diagnosis of patients with deep infiltrative endometriosis in comparison with intraoperative findings to confirm the diagnosis .

CONTACTS AND LOCATIONS:
Locations (1):
- Alexandria Faculty Of Medicine, Alexandria, El Shatby, Egypt